CLINICAL TRIAL: NCT01878682
Title: A Study to Evaluate the Performance of the VibraTip® Product by Different Community Medical Practitioners Compared to an Expert Validation by a Diabetologists.
Brief Title: A Study to Evaluate the Performance of VibraTip® by Different Clinical Users
Status: Completed | Type: Observational
Sponsor: Tameside Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Edward Jude, Consultant Physician, Tameside Hospital NHS Foundation Trust
Other Study IDs: VibraTip® SSFHC/002
Record Dates: First submitted 2013-06-08; First posted 2013-06-17 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
VibraTip® is a pocket-sized, wipe-clean, disposable device that provides a consistent source of gentle vibration. It has been specifically designed to overcome the limitations of tuning forks for testing the integrity of vibration sense in clinic and by the bedside. The product is a hand held device that is used to examine the feet of Diabetic patients who are susceptible to peripheral neuropathy that can in turn lead to ulcers. Treatment is expensive and can be over a period of time, often not being completely resolved, and can lead to amputation. The product will increase awareness of foot care and achieve a reduction in incidence of foot ulcers.

The study aims to evaluate the accuracy of the VibraTip device compared to the Gold Standard, the 10g Semmes Weinstein Monofilament (MF) Test, and the accuracy and usability of the VibraTip® device, as measured by different community medical practitioners.

DETAILED DESCRIPTION:
Primary Objective The accuracy of the VibraTip® device, as measured by a comparison with the Gold Standard, the 10g Semmes Weinstein Monofilament (MF) Test by a Diabetologist.

Secondary Objectives The accuracy and usability of the VibraTip® device, as measured by different community medical practitioners compared to expert validation by a Diabetologist.

Prospective, single centre diagnostic evaluation. A single centre in the UK (Tameside Hospital NHS Foundation Trust). Patients will be recruited while attending Tameside Hospital NHS Foundation Trust Diabetes Clinic for a routine 12 month diabetes check up. Subjects will receive a Patient Letter to invite them to take part in the VibraTip study and a Patient Information Leaflet about the study enclosed within their Diabetes Clinic appointment. The study will aim to invite 180 patients to take part in the study and aims to recruit 100 subjects into the study within 3 months. Subjects aged 18 to 75 (inclusive) of either sex with pre-existing diabetes (Type 1 and Type 2). The study aims to recruit approximately 50 (50%) of patients with diabetic peripheral neuropathy (both painful and painless) and 50 (50%) without diabetic peripheral neuropathy. (we will go for even split if possible)

ELIGIBILITY:
Inclusion Criteria:

Subjects aged 18 to 75 (inclusive) of either sex Subjects from whom consent has been obtained Subjects with pre-existing diabetes (Type 1 and Type 2)

Exclusion Criteria:

* Subjects unable to give consent
* Subjects aged less than 18 years or over 75 years
* Subjects with non-diabetic causes of neuropathy
* Subjects who have already taken part in the study
* Subjects who have active foot ulceration on the big toe
* Subjects who have PAD ABPI < 0.7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited while attending Tameside Hospital NHS Foundation Trust Diabetes Clinic for a routine 12 month diabetes check up
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2014-07-10 (Actual)

PRIMARY OUTCOMES:
The accuracy of the VibraTip® device, as measured by a comparison with the Gold Standard, the 10g Semmes Weinstein Monofilament (MF) Test by a Diabetologist. | 3 months
  The accuracy of the VibraTip® device, as measured by a comparison with the Gold Standard, the 10g Semmes Weinstein Monofilament (MF) Test by a Diabetologist.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Jude, MD, Principal Investigator — Tameside Hospital NHS Foundation Trust
Locations (1):
- Tameside Hospital NHS Foundation Trust, Ashton-under-Lyne, Lancs, United Kingdom